CLINICAL TRIAL: NCT04178239
Title: Neuropsychobiological Fingerprints of Chronic Fatigue in Sarcoidosis
Brief Title: Chronic Fatigue in Sarcoidosis
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Michael Dreher, Univ.-Prof. Dr. med. Michael Dreher, RWTH Aachen University
Other Study IDs: 16-082
Record Dates: First submitted 2019-11-18; First posted 2019-11-26 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Sarcoidosis
Keywords: Fatigue; fMRI
MeSH Terms: conditions — Sarcoidosis; Fatigue | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Fatigue: MFI score >53 points
  Interventions: Diagnostic Test: fMRI, questionnaires, pneumologic diagnostics
- No Chronic Fatigue: MFI score < 54 points
  Interventions: Diagnostic Test: fMRI, questionnaires, pneumologic diagnostics

INTERVENTIONS:
Diagnostic Test: fMRI, questionnaires, pneumologic diagnostics — fMRI neuropsychological questionnaires pneumologic diagnostics: blood samples, whole body plethysmography, walking test

SUMMARY:
Background: Chronic fatigue (CF) is a prominent symptom in many sarcoidosis patients, affecting quality of life (QoL) and interfering with treatment. This study investigates neuropsychobiological mechanisms and markers of CF in sarcoidosis.

DETAILED DESCRIPTION:
Patients with a histological diagnosis of sarcoidosis are included. The Multidimensional Fatigue Inventory (MFI) is used to define patients with and without CF. All patients are then characterized using several fatigue, depression, QoL and executive functioning questionnaires. Cognitive functioning and underlying neural correlates are assessed using an n-back task measuring working memory and (sustained) attention during functional magnetic resonance imaging (fMRI). Sarcoidosis disease activity is determined using lung function, laboratory parameters, and exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* histologically diagnosed sarcoidosis
* age ≥18 years
* provision of written informed consent
* sufficient German language skills to fully understand all questionnaires

Exclusion Criteria:

* patients unable to understand study-related information
* insufficient language skills in German language
* MRI-related contraindications:
* any kind of implants or extraneous material inside the body
* past thoracic or ophthalmologic surgery
* medical history of epilepsy, tinnitus or seizure
* extensive tattoos
* current pregnancy
* claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sarcoidosis patients (histologically diagnosed)
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity | 1 day of study participation
  Measured by a Fatigue questionnaire that has frequently been used in cohorts of sarcoidosis patients, the Multidimensional Fatigue Inventory (MFI).
  It consists of 20 items. For each item a score of 1 to 5 is possible, resulting in a total score of 20-100. Higher scores indicate a higher level of fatigue. In this study fatigue is diagnosed in patients with a total score of >53 based on the 75th percentile of norm values as primary developed by Kuhnt et al and used in several studies with cohorts of sarcoidosis patients.
Fatigue | 1 day of study participation
  In addition to the MFI the Fatigue Assessement Scale (FAS) is performed. It is frequently used in cohorts of sarcoidosis patients. With its 10 Items the possible total score varies from 10 to 50, higher scores indicate more fatigue.
Impact of fatigue on health-related quality of life | 1 day of study participation
  Assessed by the Fatigue Impact Scale (FIS). It includes 40 items resulting in a total score from 0 to 160. Higher values indicate more fatigue.
Cognitive functioning and underlying neural correlates | 1 day of study participation
  Assessed by an n-back task measuring working memory and (sustained) attention during functional magnetic resonance imaging.
  Reaction times and hit rates are measured.
Sarcoidosis disease activity | 1 day of study participation
  Is assessed by s-IL2-receptor (U/ml), ACE-polymorphism (mU/L) and Neopterin (nmol/L) values from a blood sample. Higher values indicate a higher sarcoidosis disease activity.
Lung function assessement | 1 day of study participation
  Whole body plethysmography is performed according to current recommendations. Parameters measured include total lung capacity (% predicted), vital capacity (% predicted), FEV1 (% predicted) and DLCO (% predicted).
Exercise Capacity | 1 day of study participation
  Assessed by a standardised six-minute walking test. Walking distance the patient achieves within six minutes is assessed.
Quality of life (self-assessment) | 1 day of study participation
  Assessed by the World Health Organization quality of Life Questionnaire, short form (WHO-QOL-BREF). The included Items assess aspects of quality of life in different domains: physical health domain, psychologic health domain, social relationships domain, environmental health domain, global domain. Domain scores are scaled in a positive direction, therefore higher scores denote higher quality of life. Scores from 0 to 100 are possible in each domain.
Depression (self-assessment) | 1 day of study participation
  Patients are asked to perform the ADS (Allgemeine Depressionsskala). A total score from 0 to 60 points is possible, while higher scores indicate more signs and symptoms of depression.
Depression (third-party-assessment) | 1 day of study participation
  Assessed by the Hamilton Depression Scale (HAMD). A total score of 0 to 62 points is possible with higher scores indicating more signs and symptoms of depression.
Anxiety | 1 day of study participation
  Assessed by the State-Trait-Anxiety-Inventory (STAI). It consists of two subscales, each including 20 items. For each subscale there is a possible score from 20 to 80 points with higher scores indicating more anxiety.
Executive functioning | 1 day of study participation.
  Assessed by the Trail-Making-Test (TMT-A and -B). Time necessary for completion of the task is measured, shorter periods of time indicate a better executive functioning in terms of attention.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Principal Investigator — RWTH Aachen University Hospital
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Kettenbach S, Radke S, Muller T, Habel U, Dreher M. Neuropsychobiological Fingerprints of Chronic Fatigue in Sarcoidosis. Front Behav Neurosci. 2021 Jul 26;15:633005. doi: 10.3389/fnbeh.2021.633005. eCollection 2021. PMID 34381339